CLINICAL TRIAL: NCT02472561
Title: Verizon mHealth Solution for Elderly Underserved Patients With Peripheral Artery Disease
Brief Title: Verizon mHealth Solution for Patients With Peripheral Artery Disease (PAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Verizon Wireless (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00059885
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Peripheral Artery Disease
Keywords: Cardiology; Vascular; Peripheral Artery Disease; Artery; Mobile Health; Exercise; PAD
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobile Health Application Group 1 (Experimental): Participants will wear a Fitbit Physical Activity Monitor to objectively quantify physical activity patterns. Once a week (± 3 days) during the 12 week mHealth intervention patients will measure and download their blood pressure and blood glucose (if diabetic) by means of a mHealth blood pressure cuff and mHealth glucometer. Medication adherence will be measured at baseline and 12-weeks by the Morisky Medication Adherence Scale-8 (MMAS-8) questionnaire. Each participant will be provided with a electronic version of the book titled, "Your COMPLETE and EASY GUIDE to Understanding Peripheral Artery Disease"; patients will be asked to read approximately one chapter per week for educational purposes.
  Interventions: Other: Fitbit Physical Activity Monitor; Other: mHealth Glucometer; Other: mHealth Blood Pressure
- Usual Care Group 2 (No Intervention): Participants will follow standard care as ordered by their individual, treating physician. Each participant will be given a paperback copy of the book, "Your COMPLETE and EASY GUIDE to Understanding Peripheral Artery Disease". All participants will be contacted by study personnel in order to schedule visits at baseline and 12-weeks for the outcome assessments.

INTERVENTIONS:
Other: Fitbit Physical Activity Monitor — Physical Activity: The study team will provide an individualized goal of total number of steps to attain daily and will be monitored using a Fitbit activity tracker. The total daily step goal will be reviewed by study staff and modified at weeks 4 and 8.
  Arms: Mobile Health Application Group 1
Other: mHealth Glucometer — Blood Glucose: The participant will monitor their fasting blood glucose once per week by using an mHealth Glucometer and mobile app.
  Other Names: Diabetics Only
  Arms: Mobile Health Application Group 1
Other: mHealth Blood Pressure — Blood Pressure: The participant will monitor their blood pressure once per week by using an mHealth Blood Pressure cuff and mobile app.
  Arms: Mobile Health Application Group 1

SUMMARY:
The purpose of this study is to understand the effects that a three month lifestyle-based mobile health (mHealth) peripheral artery disease (PAD) prevention program will have on improving physical activity, fitness, important PAD risk factors and quality of life (QOL) in patients with PAD.

By testing a novel mHealth intervention focused on lifestyle modification, this trial will address a critical evidence gap in the care of PAD patients. PAD patients are not eligible for cardiac rehabilitation and therefore struggle with unhealthy lifestyles, and these patients currently have no lifestyle-based care strategies to help them. The results of this study have the potential to lead to new sustainable and resource-efficient, lifestyle-based preventive care strategies for patients with stable PAD.

DETAILED DESCRIPTION:
This is a single-center, randomized trial designed to examine the hypothesis that a lifestyle-based mHealth peripheral artery disease (PAD) prevention program will improve physical activity, fitness, important PAD risk factors and quality of life (QOL).

The investigators may enroll up to 55 men and women being evaluated for leg pain from Duke PAD cardiovascular clinics or after lower extremity angioplasty in the Duke catheterization laboratory. Of the 55 men and women volunteers who may be initially consented, the investigators anticipate a portion (potentially 20%) may drop out during the study timeline, and approximately 45 are expected to complete this study. Following informed consent and baseline testing, the participants will be randomized (1.25:1.00) into either a mHealth (N=25) or usual care group (N=20) [for comparison] for a 12-week period. All patients will be evaluated for walking ability on a treadmill test, quality of life questionnaires, health literacy related to PAD and the most important risk factors specific to PAD (blood glucose if diabetic, daily physical activity and blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* Adequate clinical stability has been achieved in the judgment of the investigator to allow participation in study assessments and the intervention
* A history of stable intermittent claudication for >2 months, and an ABI <0.9 at rest
* No contraindications to exercise training
* All subjects will be on the recommended regimen of statin and antiplatelet therapy
* Signed informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study

Exclusion Criteria:

* Present or a past history of gangrene, impending limb loss or osteomyelitis
* Severe peripheral neuropathy
* Any condition other than PAD that limits walking for example arthritis or chronic obstructive pulmonary disease (COPD)
* Unstable angina, history of significant left main disease or three vessel coronary artery disease (>70% stenosis, unprotected by grafts) or recent myocardial infarction (less than eight weeks)
* Chest pain during treadmill exercise which appears before the onset of claudication, or 2 mm ST depression during exercise regardless of the results of tests for myocardial ischemia
* Refusal or inability to give informed consent or inability or unwillingness to comply with the study requirements.
* Dementia that precludes ability to participate in and follow study protocols
* Enrollment in a clinical trial not approved for co-enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular fitness level measured by change score analysis of peak Volume of Oxygen (pVO2mL/kg/min) consumption measured during a cardiopulmonary exercise test (CPET). | Baseline and 12-week
  peak VO2 mL/kg/min

SECONDARY OUTCOMES:
Feasibility of this novel mobile health treatment strategy, as measured by patient satisfaction survey | 12-week
  Patient Satisfaction Survey
Implementation of this novel mobile health treatment strategy, as measured by patient satisfaction | 12-week
  Patient Satisfaction Survey
Change in physical activity patterns (steps, time and distance) | Baseline and 12-week
  Steps, time and distance per week
Change score analysis in Body Mass Index measurements | Baseline and 12-week
  Ratio of height to weight
Change score analysis in Blood Glucose measurements | Baseline and 12-week
  Fasting Plasma Glucose and Hemoglobin A1-C
Change in Medication Adherence scores as measured by the Morisky Medication Adherence Scale (MMAS-8) | Baseline and 12-week
Change in Quality of Life (QOL) scores on the Walking Impairment Questionnaire | Baseline and 12-week
Change in Peripheral Artery Disease (PAD) Health Aptitude scores on the Health Aptitude Questionnaire | Baseline and 12-week
Change in Smoking Habits scores on the PAD: Smoking Habit Questionnaire | Baseline and 12-week
Change score analysis in Systolic and Diastolic Blood Pressure measurements | Baseline and 12-week

CONTACTS AND LOCATIONS:
Overall Officials: Manesh R Patel, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States